CLINICAL TRIAL: NCT01560000
Title: Effect of Bran Fiber Type on Subjective and Objective Measures of Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1202E10321
Record Dates: First submitted 2012-03-05; First posted 2012-03-21 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Food
Keywords: The focus of this study is to determine satiety
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- fiber (Other)
  Interventions: Dietary Supplement: Dietary fiber

INTERVENTIONS:
Dietary Supplement: Dietary fiber — Wheat, barley, oat and bran fibers added to a breakfast product

SUMMARY:
The objective of this study is to determine the satiety value of different bran fibers on appetite & subsequent food intake with acute consumption. Satiety will be measured subjectively by visual analogue scales (VAS).

DETAILED DESCRIPTION:
Visual analogue scales will be used to measure satiety at 15, 30 45, 60, 120, 180, and 240 minutes

ELIGIBILITY:
Inclusion Criteria:

* healthy women between the ages of 18-40
* body mass index between 18.5-29.9kg/m2
* eat breakfast regularly
* nonsmoking
* not taking weight loss medications
* non-dieting (weight stable over the past 3 months)
* spoken and written English literacy.

Exclusion Criteria:

* antibiotic use within the past 6 months
* cardiovascular disease
* diabetes mellitus
* cancer in the past 5 years
* renal or hepatic disease
* recent bacterial infection
* gastrointestinal conditions affecting digestion or absorption
* weight loss>5kg in prior 3 months (intentional or unintentional)
* history of drug or alcohol abuse in prior 6 months
* food allergies
* high fiber intake(3 or more servings of high fiber foods per day)
* lipid-lowering, anti-hypertensive or anti-inflammatory steroid medication use
* restrained eater(score>10 on the dietary restraint factor of the Three Factor Eating Questionnaire)
* concurrent or recent (within 30 days) participation in an intervention study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Satiety response | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Korczak R, Lindeman K, Thomas W, Slavin JL. Bran fibers and satiety in women who do not exhibit restrained eating. Appetite. 2014 Sep;80:257-63. doi: 10.1016/j.appet.2014.05.025. Epub 2014 May 27. PMID 24874565